CLINICAL TRIAL: NCT04055727
Title: Sepsis at Södersjukhuset-Adherence to Treatment Guidelines
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Katarina Bohm, Associate Professor, Karolinska Institutet
Other Study IDs: SepsisSoS
Record Dates: First submitted 2019-08-12; First posted 2019-08-14 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Sepsis
Keywords: treatment
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A retrospective single-center study with patients with suspected sepsis admitted to the Emergency Department at Södersjukhuset during a period of two years. The aim is to describe the association between adherence to treatment guidelines, gender, incidence and mortality for patients with sepsis.

DETAILED DESCRIPTION:
In this single-center study, patients with suspected sepsis admitted to the Emergency Department at Södersjukhuset during a period of two years will be included. About 11,000 patients will be included. Patient data including described sepsis symptoms will be drawn from the electronic medical record, TakeCare and Clinisoft. Logistic regression analysis will adjust for age, gender, comorbidity according to Charlson score, vital signs, with preliminary focus of infection (pneumonia, urinary tract infection, abdominal, other, unknown). The Surviving Sepsis guidelines for the time period are: 3-hour bundle including lactate measurement, obtaining blood culture, fluid treatment if hypotensive and administration of broad-spectrum antibiotics. The 6-hour bundles with administration of vasopressors if needed, remeasure lactate if elevated, with persistent hypotension re-asses volume status and tissue perfusion. Time zero is defined as the admission time to the emergency department. The aim is to describe the association between adherence to treatment guidelines, gender, incidence and mortality for patients with sepsis.

ELIGIBILITY:
Inclusion criteria:

• Patients admitted to the Emergency Department at Södersjukhuset with suspicion of sepsis defined as blood cultures taken and intravenous antibiotics of type beta-lactam or aminoglycoside prescribed within 48 hours of admission.

Exclusion criteria:

• Patients transferred from other hospitals or treatment clinics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the emergency department at Södersjukhuset
Sampling Method: Probability Sample
Enrollment: 11000 (Estimated)
Dates: Start 2019-03-07 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Gender differences in 90-day mortality | 90 days
  Gender differences in percentage of patients who died before day 90

SECONDARY OUTCOMES:
Association between adherence to treatment guidelines and mortality | 90 days
  Association between number of completed sepsis bundles and mortality
Incidence of sepsis | 90 days
  Number of patients admitted to the Emergency Department at Södersjukhuset during the study period comparing to the hospitals catchment area

CONTACTS AND LOCATIONS:
Overall Officials: Katarina Bohm, Ass Prof, Principal Investigator — Karolinska Institutet
Locations (1):
- Södersjukhuset, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No